CLINICAL TRIAL: NCT01193777
Title: L-Carnitine Administration in Early Sepsis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped to open expanded phase II study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-10-06A; 10POST3560001 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2010-08-30; First posted 2010-09-02 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2012-03

CONDITIONS: Septic Shock
Keywords: Carnitine; Shock; Sepsis
MeSH Terms: conditions — Shock, Septic; Shock; Sepsis | interventions — Carnitine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline
- L-Carnitine (Experimental)
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine — 4 gram bolus followed by 8 gram in 1 L NS infused over 12 hours.
  Arms: L-Carnitine
Drug: Normal Saline — Bolus followed by 1 L NS infusion over 12 hours.
  Arms: Saline

SUMMARY:
Sepsis is a severe and overwhelming response to an infection in the body. Over 750,000 patients in the United States develop sepsis every year. As sepsis becomes progressively more severe, a patient's blood pressure drops to dangerous levels and the body cannot pump oxygen to the rest of the body, which is necessary for normal cell function. This is called septic shock. When someone develops septic shock, it is very common for the smallest blood vessels in the body called the microcirculation to clog, like a highway during rush hour. Even with the best medical care, more than one in three patients with septic shock will die.

The major goal of this study is to test if intravenous replacement of a naturally occurring nutrient that is lost by the body during sepsis called L-carnitine can reduce how sick a patient with sepsis becomes. In our study, some patients will receive L-carnitine and others will receive saline. We will measure markers determining severity of illness in both groups and compare them to see if L-carnitine helps patients get better faster. Based on research already conducted, we believe L-carnitine will improve blood flow in the microcirculation, delivering more oxygen to cells, and help the body get better. To test if this is true, we will directly look at the microcirculation under the tongue with a special magnifying camera that looks at red blood cells, and compare both groups.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection
* Any two of four criteria of systemic inflammatory response
* Requirement for vasopressors to treat shock
* Enrollment within 12 hours of vasopressor initiation
* SOFA score of greater than or equal to 5 at the time of enrollment

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* Any primary diagnosis other than sepsis
* Established Do Not Resuscitate status or advanced directives restricting aggressive care or treating physician deems aggressive care unsuitable
* Any history of seizures or a known seizure disorder
* Any known inborn error of metabolism
* Anticipated requirement for surgery that would interfere with the 12 hour infusion time
* Active participation in another interventional study
* Inability to obtain informed consent
* Cardiopulmonary resuscitation (chest compression or defibrillation) prior to enrollment
* Known systemic allergy to carnitine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in organ failure | 24 hours
  SOFA score will be measured at 0 and 24 hours

SECONDARY OUTCOMES:
Microcirculation | 12 hours
  Test if carnitine improves blood flow in the sublingual microvasculature during septic shock by performing sidestream dark-field (SDF) video-microscopy of the sublingual microcirculation, prior to and after 12 hours of carnitine infusion.
ICU and hospital length of stay | Duration of stay
All-cause mortality | 28 day
All-cause mortality | 3 months
All-cause mortality | 6 months
All-cause mortality | 12 months
Change in inflammatory markers | 12 hours
  Assess change in various inflammatory markers over predefined time points.
Change in inflammatory markers | 24 hours
  Assess change in various inflammatory markers over predefined time points.
Change in inflammatory markers | 48 hours
  Assess change in various inflammatory markers over predefined time points.

CONTACTS AND LOCATIONS:
Overall Officials: Alan E Jones, MD, Principal Investigator — University of Mississippi and Carolinas Medical Center, Department of Emergency Medicine
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Carolinas Medical Center, Charlotte, North Carolina

REFERENCES:
- [Derived] Puskarich MA, Shapiro NI, Massey MJ, Kline JA, Jones AE. Lactate Clearance in Septic Shock Is Not a Surrogate for Improved Microcirculatory Flow. Acad Emerg Med. 2016 Jun;23(6):690-3. doi: 10.1111/acem.12928. Epub 2016 May 11. PMID 26825368